CLINICAL TRIAL: NCT05314595
Title: The Effect of Bilateral Uterine Artery Ligation as an Added Step for Placental Pouch Closure Technique in Management of Placenta Accreta Spectrum on Reducing Intra-operative Blood Loss: A Comparative Study
Brief Title: Bilateral Uterine Artery Ligation in PPC Technique for Management of PAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Hussein Abouzeid Ahmed, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAS
Record Dates: First submitted 2022-03-11; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- modified technique (Experimental): women were underwent modified technique (PPC+ bilateral uterine artery ligation)
  Interventions: Procedure: bilateral uterine artery ligation

INTERVENTIONS:
Procedure: bilateral uterine artery ligation — * Spinal anaethesia with intrathecal morphia
  * Transverse skin incision
  * Adequate dissection of the bladder.
  * Incision of the uterus above placental edge.
  * Delivery of the fetus.
  * Delayed cord clamping (60 seconds) if the baby appears well.
  * Exteriorization of the uterus.
  * Start Oxytocin infusion and uterine massage to ensure good uterine contractions immediately after delivery of the fetus. No trials of placental delivery will be made at this point.
  * At this point, a gentile trial to deliver the placenta is performed
  * A catheter is placed in the cervix from above to secure the cervical opening
  * Compression is applied to the site of bleeding from placenta site
  * Placental pouch is marked by multiple allies and is closed down to the multiple-8 suture.
  * Blood loss is measured using the suction device and coated socked towels. In modified PPC, Bilateral uterine artery ligation will be done after exteriorization of the uterus in order to minimize the blood loss.

SUMMARY:
Aim of the study

Primary outcomes:

1. The effect of bilateral uterine artery ligation in reducing intraoperative bleeding in women underwent PPC as a conservative surgical technique.
2. Decrease surgical time.

Secondary outcomes:

1. Associated maternal morbidity and mortality.
2. Amount of blood transfusion
3. Difference in hematocrit value before and after delivery

DETAILED DESCRIPTION:
Introduction Placenta accreta spectrum (PAS) is a term that comprises abnormal placental invasion disorders of the uterine wall. According to the depth of invasion, it ranges from placental invasion in contact with myometrium (placenta accreta), into myometrium (placenta increta), or beyond myometrium (placenta percreta) (Tan, Tay et al. 2007, Cal, Ayres-de-Campos et al. 2018). PAS is an obstetric emergency that may be complicated by emergency hysterectomy, intraoperative surgical complications, massive transfusion, hemorrhagic shock, and even maternal death if not managed efficiently (Ye 2017). Previous cesarean deliveries, placenta previa and advanced maternal age are recognized strong risk factors of PAS, all of which, have become more prevalent among contemporary population (Silver, Landon et al. 2006, Zeng, Yang et al. 2018). Therefore, PAS is no longer a rare disorder in modern practice; the incidence of PAS has increased from approximately 1 in 30,000 deliveries before 1950 to 3 in 1000 deliveries in the current decade (Timor-Tritsch, Monteagudo et al. 2012).

Currently, cesarean hysterectomy is the standard management of PAS (Matsubara, Kuwata et al. 2013). Despite surgical risks, loss of uterine function, and psychological sequences, cesarean hysterectomy permits elective intervention under controlled settings to minimize blood loss (2002). Although several uterus-conserving interventions have been proposed in management of PAS, their contribution to evidence-based practice is limited (Jauniaux, Alfirevic et al. 2018), and cesarean hysterectomy is endorsed as the standard intervention (gynaecology, Gynaecology et al. 2002). Cesarean hysterectomy, without attempting to remove the placenta, may reduce risk of significant bleeding and associated morbidity (Eller, Porter et al. 2009). Leaving the placenta in situ is endorsed as an alternative in patients who refuse hysterectomy being the least invasive uterus-conserving intervention (Jauniaux, Alfirevic et al. 2018, Sentilhes, Kayem et al. 2018).

Nevertheless, the need for evidence-based conservative approaches for PAS cannot be underestimated particularly among women who are highly motivated to preserve their fertility. Despite limited evidence, an international survey indicates that 39% of obstetricians consider conservative management as the primary management. Notably, conservative management was inconsistent among respondents (Cal, Ayres-de-Campos et al. 2018).

Placental pouch closure looks to be an attractive and effective surgical procedure for conservative management of placenta accreta (Zahran, Elsonbaty et al. 2020). In their series of 60 Placenta accreta cases reported that by using this technique,59 out of the 60 enrolled cases, the uterus was successfully conserved and there were no cases of maternal mortality or severe morbidities related to the procedure.

Major blood supply of the uterus comes from the uterine artery, so bilateral uterine artery ligation (UAL) before delivering of the placenta greatly decreasing the blood loss(Lin, Lin et al. 2019). Simultaneously, the ovarian blood flow has not been affected and consequently no changes in ovarian reserve markers occurred, so it is considered one of preserving fertility surgical technique (Verit, Çetin et al. 2019).

ELIGIBILITY:
Inclusion Criteria:

* • Previous operations

  * Gestational age (28 weeks)
  * Prenatally suspected PAS based on sonographic and/or MRI findings and/or intrapartum diagnosis of PAS.
  * Authorization to participate in the study

Exclusion Criteria:

* • Coagulopathies

  * Chronic renal or hepatic impairment (baseline first trimester labs are beyond normal range for pregnancy)
  * Delivery in an outside hospital (patients referred for ongoing massive bleeding due to PAS)
  * Patients coming in emergency condition with bleeding or in labour.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
bilateral uterine artery ligation | 30 months
  1. The effect of bilateral uterine artery ligation and estimation of blood volume loss (VMBL): direct measurement of blood loss in volume units (mL);

CONTACTS AND LOCATIONS:
Overall Officials: Kamal M Zahran, Professor, Study Chair — Assiut medical school
Locations (1):
- Assiut Medical School, Asyut, Egypt

REFERENCES:
- [Background] Cal M, Ayres-de-Campos D, Jauniaux E. International survey of practices used in the diagnosis and management of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2018 Mar;140(3):307-311. doi: 10.1002/ijgo.12391. Epub 2017 Dec 22. PMID 29149470
- [Background] Tan CH, Tay KH, Sheah K, Kwek K, Wong K, Tan HK, Tan BS. Perioperative endovascular internal iliac artery occlusion balloon placement in management of placenta accreta. AJR Am J Roentgenol. 2007 Nov;189(5):1158-63. doi: 10.2214/AJR.07.2417. PMID 17954654
- [Background] Ye M, Yin Z, Xue M, Deng X. High-intensity focused ultrasound combined with hysteroscopic resection for the treatment of placenta accreta. BJOG. 2017 Aug;124(Suppl 3):71-77. doi: 10.1111/1471-0528.14743. PMID 28856861
- [Background] Silver RM, Landon MB, Rouse DJ, Leveno KJ, Spong CY, Thom EA, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal morbidity associated with multiple repeat cesarean deliveries. Obstet Gynecol. 2006 Jun;107(6):1226-32. doi: 10.1097/01.AOG.0000219750.79480.84. PMID 16738145
- See also: International survey of practices used in the diagnosis and management of placenta accreta spectrum disorders — https://pubmed.ncbi.nlm.nih.gov/29149470/
- See also: Perioperative endovascular internal iliac artery occlusion balloon placement in management of placenta accreta — https://pubmed.ncbi.nlm.nih.gov/17954654/
- See also: High-intensity focused ultrasound combined with hysteroscopic resection for the treatment of placenta accreta — https://pubmed.ncbi.nlm.nih.gov/28856861/
- See also: Placenta accreta spectrum disorder trends in the context of the universal two-child policy in China and the risk of hysterectomy — https://pubmed.ncbi.nlm.nih.gov/29214633/
- See also: Maternal morbidity associated with multiple repeat cesarean deliveries — https://pubmed.ncbi.nlm.nih.gov/16738145/
- See also: Unforeseen consequences of the increasing rate of cesarean deliveries: early placenta accreta and cesarean scar pregnancy. A review — https://pubmed.ncbi.nlm.nih.gov/22516620/